CLINICAL TRIAL: NCT06153485
Title: Effectiveness of Automated Titration Designed for Home Oxygen Therapy
Brief Title: Automated Titration for Home Oxygen Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Director, Program in Respiratory Rehabilitation, West Park Healthcare Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AutoO2x
Record Dates: First submitted 2023-11-02; First posted 2023-12-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Chronic Respiratory Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AutoO2 (Experimental): Automated Titration of Oxygen (Auto-O2) using a closed-loop system in which the oxygen flow to the participant is continuously adjusted on the basis of pulse oximetry signals to maintain a target range of oxygen saturation to meet the patient's immediate needs.
  Interventions: Device: AutoO2
- FixedO2 (Active Comparator): Fixed flow oxygen delivery administered using manual flow meters according to standard clinical procedures.
  Interventions: Other: FixedO2

INTERVENTIONS:
Device: AutoO2 — Automated Titration of Oxygen (Auto-O2) using a closed-loop system in which the oxygen flow to the participant is continuously adjusted on the basis of pulse oximetry signals to maintain a target range of oxygen saturation to meet the participant's immediate needs.
  Other Names: HOT-100 (O2matic Ltd, Herlev, Denmark)
  Arms: AutoO2
Other: FixedO2 — Fixed flow oxygen delivery administered using manual flow meters according to standard clinical procedures.
  Arms: FixedO2

SUMMARY:
Patients with chronic respiratory disease may be prescribed oxygen therapy. Currently, the dose of oxygen flow is fixed (FixedO2) depending on activity level i.e. rest, physical activity and sleep. Automated Titration of Oxygen (AutoO2) is a closed-loop system in which the oxygen flow to the patient is continuously machine adjusted to meet the patient's immediate needs on the basis of signals from pulse oximetry (SpO2). The purpose of this study is to examine if automated oxygen control based on pulse oximetry provided to participants is superior to prescribed fixed oxygen flow in keeping SpO2 within the intended target interval of 92 to 96% arterial oxygen saturation.

DETAILED DESCRIPTION:
Patients with chronic respiratory disease may be prescribed oxygen therapy. Currently, the dose of oxygen flow is fixed (FixedO2). The fixed flow is adjusted by category of activity (rest, physical activity and sleep) hereafter known as their state. The flow remains the same throughout each state and day-to-day regardless of the patient's disease status. Automated Titration of Oxygen (AutoO2) is a closed-loop system in which the oxygen flow to the patient is continuously machine adjusted to meet the patient's immediate needs on the basis of signals from pulse oximetry (SpO2). The auto-titration system used in this study is intended for home use by patients for whom home oxygen has been prescribed. It includes the central monitoring of automatic titration. Before its use at home, it must demonstrate its abilities consistently in a supervised free living environment. In this crossover trial patients already using supplemental oxygen and admitted to one of West Park Healthcare Centre's in-patient respiratory programs are exposed to alternating consecutive weeks of: 1) usual fixed dose oxygen, or; 2) automated oxygen titration. The purpose of this study is to examine if automated oxygen control based on pulse oximetry provided to participants is superior to prescribed fixed oxygen flow in keeping SpO2 within the intended target interval. To determine whether AutoO2 provides a more precise method of supplemental oxygen delivery manifested by greater amount of time within a targeted oxygen saturation (%t92-96) compared to fixed flow oxygen therapy in individuals with chronic respiratory disease. Participants will be randomised 1:1 to start with FixedO2 or AutoO2 using a computer generated block randomisation scheme. They will then alternate between conditions weekly over 4 weeks. Participants will use their usual oxygen delivery method and equipment. The AutoO2 will be inserted in-line as part of the participant's usual fixed flow system. All patient activities associated with their participation in the pulmonary rehabilitation program are unchanged. We will use continuous activity monitoring to categorize activity state i.e.rest, physical activity or sleep. Cardiac pulse from the oximeter will be used to corroborate the activity state. We will record oxygen flow from the source to the participant.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic respiratory disease
* current prescription for supplemental oxygen therapy

Exclusion Criteria:

* characteristics that compromise the validity of oximetry
* inability to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily time spent normoxic as defined by an arterial oxygen saturation measured by pulse oximetry (SpO2), between 92 to 96%, will be expressed a function of total time recorded SpO2. | 24 hour
  SpO2 will be recorded throughout the day (24 hours). The primary outcome measure equals the daily time with 92%≥SpO2≤ 96% (numerator) divided by the total daily time of measured SpO2 (denominator).

CONTACTS AND LOCATIONS:
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No